CLINICAL TRIAL: NCT00098306
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of a Novel CCR5 Antagonist, UK-427,857, in Combination With Optimized Background Therapy Versus Optimized Background Therapy Alone for the Treatment of Antiretroviral-Experienced HIV-1 Infected Subjects.
Brief Title: Trial of Maraviroc (UK-427,857) in Combination With Optimized Background Therapy Versus Optimized Background Therapy Alone for the Treatment of HIV-1 Infected Subjects
Acronym: MOTIVATE 1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A4001027
Record Dates: First submitted 2004-12-06; First posted 2004-12-07 (Estimated); Results first posted 2012-04-27 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Maraviroc (UK-427,857); Drug: Optimized Background Therapy
- 2 (Experimental)
  Interventions: Drug: Optimized Background Therapy; Drug: Placebo
- 3 (Experimental)
  Interventions: Drug: Optimized Background Therapy

INTERVENTIONS:
Drug: Maraviroc (UK-427,857) — Maraviroc was given either once or twice per day with the dose adjusted according to the optimized background therapy
  Other Names: Selzentry
  Arms: 1
Drug: Optimized Background Therapy — Maraviroc was given either once or twice per day with the dose adjusted according to the optimized background therapy
  Arms: 1
Drug: Optimized Background Therapy — Patients will be randomly (2:2:1) assigned to one of three groups: Optimized Background Therapy [OBT (3-6 drugs based on treatment history and resistance testing)] + maraviroc (UK-427,857) 150 mg taken once daily, OBT + maraviroc (UK-427,857) 150 mg taken twice daily, or OBT alone.
  Arms: 2
Drug: Placebo — Patients will be randomly (2:2:1) assigned to one of three groups: Optimized Background Therapy [OBT (3-6 drugs based on treatment history and resistance testing)] + maraviroc (UK-427,857) 150 mg taken once daily, OBT + maraviroc (UK-427,857) 150 mg taken twice daily, or OBT alone.
  Arms: 2
Drug: Optimized Background Therapy — Patients will be randomly (2:2:1) assigned to one of three groups: Optimized Background Therapy [OBT (3-6 drugs based on treatment history and resistance testing)] + maraviroc (UK-427,857) 150 mg taken once daily, OBT + maraviroc (UK-427,857) 150 mg taken twice daily, or OBT alone. The study will enroll over approximately a 9 month period with 48 weeks of treatment.
  Arms: 3

SUMMARY:
Maraviroc (UK-427,857), a selective and reversible CCR5 coreceptor antagonist, has been shown to be active in vitro against a wide range of clinical isolates (including those resistant to existing classes). In HIV-1 infected patients, maraviroc (UK-427,857) given as monotherapy for 10 days reduced HIV-1 viral load by up to 1.6 log, consistent with currently available agents. Safety and toleration have been studied in over 400 subjects for up to 28 days at 300 mg twice daily. No significant effects were seen on the QTc interval. The purpose of this study is to evaluate the antiretroviral activity of maraviroc (UK-427,857) in HIV infected, treatment experienced patients who are failing their current antiretroviral regimen and are infected with R5-tropic virus exclusively. This study will involve more than 100 centers from the US and Canada to achieve a total randomized subject population of 500 subjects. Patients will be randomly (2:2:1) assigned to one of three groups: Optimized Background Therapy [OBT (3-6 drugs based on treatment history and resistance testing)] + maraviroc (UK-427,857) 150 mg taken once daily, OBT + maraviroc (UK-427,857) 150 mg taken twice daily, or OBT alone. The study will enroll over approximately a 9 month period with 48 weeks of treatment. This may be extended for an additional year depending on the results at 48 weeks. Physical examinations will be performed at study entry, weeks 4, 8, 12, 16, 20, 24, 32, 40, and 48. Blood samples will also be taken at study entry, weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, and 48. Additionally, blood samples will be drawn twice, at least 30 minutes apart, at weeks 2 and 24 for maraviroc (UK-427,857) pharmacokinetic analysis. As part of this clinical study a blood sample will also be taken for non-anonymized pharmacogenetic analysis. Patients will undergo a 12-lead electrocardiogram at study entry, weeks 24 and 48.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 16 years of age (or minimum age as determined by local regulatory authorities)
* HIV-1 RNA viral load of greater than or equal to 5,000 copies/mL
* Stable pre-study antiretroviral regimen, or on no antiretroviral agents, for at least 4 weeks
* Documented genotypic or phenotypic resistance to three of the four antiretroviral drug classes, OR, Antiretroviral-class experience greater than or equal to 6 months (sequential or cumulative) with at least three of the following: One nucleoside or nucleotide reverse transcriptase inhibitor, one non-nucleoside reverse transcriptase inhibitor, two protease inhibitors (excluding low-dose ritonavir) and/or enfuvirtide
* Be willing to remain on randomized treatment without any changes or additions to the OBT regimen, except for toxicity management or upon meeting criteria for treatment failure
* A negative urine pregnancy test at the baseline visit for Women of Child Bearing Potential (WOCBP)
* Effective barrier contraception for WOCBP and males

Exclusion Criteria:

* Patients requiring treatment with more than 6 antiretroviral agents (excluding low-dose ritonavir)
* Prior treatment with maraviroc (UK-427,857) or another experimental HIV entry inhibitor for more than 14 days
* Suspected or documented active, untreated HIV-1 related opportunistic infection (OI) or other condition requiring acute therapy
* Treatment for an active opportunistic infection, or unexplained temperature >38.5 degrees Celsius for 7 consecutive days
* Active alcohol or substance abuse sufficient, in the Investigator's judgement, to prevent adherence to study medication and/or follow up
* Lactating women, or planned pregnancy during the trial period
* Significant renal insufficiency
* Previous therapy with a potentially myelosuppressive, neurotoxic, hepatoxic and/or cytotoxic agent within 30 days prior to randomization or the expected need for such therapy during the study period
* Documented or suspected acute hepatitis or pancreatitis within 30 days prior to randomization
* Significantly elevated liver enzymes or cirrhosis
* Significant neutropenia, anemia or thrombocytopenia
* Malabsorption or an inability to tolerate oral medications
* Symptomatic postural hypotension or severe cardiovascular or cerebrovascular disease
* Certain medications
* Malignancy requiring parenteral chemotherapy that must be continued for the duration of the trial
* X4- or dual/mixed-tropic virus or repeated assay failure
* Any other clinical condition that, in the Investigator's judgement, would potentially compromise study compliance or the ability to evaluate safety/efficacy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2004-11; Primary Completion 2007-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- United States (17):
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Auroa, Colorado
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Vero Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Santa Fe, New Mexico
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Annandale, Virginia
- Canada (2):
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Montreal, Quebec

REFERENCES:
- [Derived] Lewis ME, Simpson P, Mori J, Jubb B, Sullivan J, McFadyen L, van der Ryst E, Craig C, Robertson DL, Westby M. V3-Loop genotypes do not predict maraviroc susceptibility of CCR5-tropic virus or clinical response through week 48 in HIV-1-infected, treatment-experienced persons receiving optimized background regimens. Antivir Chem Chemother. 2021 Jan-Dec;29:20402066211030380. doi: 10.1177/20402066211030380. PMID 34343443
- [Derived] Gulick RM, Fatkenheuer G, Burnside R, Hardy WD, Nelson MR, Goodrich J, Mukwaya G, Portsmouth S, Heera JR. Five-year safety evaluation of maraviroc in HIV-1-infected treatment-experienced patients. J Acquir Immune Defic Syndr. 2014 Jan 1;65(1):78-81. doi: 10.1097/QAI.0b013e3182a7a97a. PMID 24419064
- [Derived] Hardy WD, Gulick RM, Mayer H, Fatkenheuer G, Nelson M, Heera J, Rajicic N, Goodrich J. Two-year safety and virologic efficacy of maraviroc in treatment-experienced patients with CCR5-tropic HIV-1 infection: 96-week combined analysis of MOTIVATE 1 and 2. J Acquir Immune Defic Syndr. 2010 Dec 15;55(5):558-64. doi: 10.1097/QAI.0b013e3181ee3d82. PMID 20703158
- [Derived] Fatkenheuer G, Nelson M, Lazzarin A, Konourina I, Hoepelman AI, Lampiris H, Hirschel B, Tebas P, Raffi F, Trottier B, Bellos N, Saag M, Cooper DA, Westby M, Tawadrous M, Sullivan JF, Ridgway C, Dunne MW, Felstead S, Mayer H, van der Ryst E; MOTIVATE 1 and MOTIVATE 2 Study Teams. Subgroup analyses of maraviroc in previously treated R5 HIV-1 infection. N Engl J Med. 2008 Oct 2;359(14):1442-55. doi: 10.1056/NEJMoa0803154. PMID 18832245
- [Derived] Gulick RM, Lalezari J, Goodrich J, Clumeck N, DeJesus E, Horban A, Nadler J, Clotet B, Karlsson A, Wohlfeiler M, Montana JB, McHale M, Sullivan J, Ridgway C, Felstead S, Dunne MW, van der Ryst E, Mayer H; MOTIVATE Study Teams. Maraviroc for previously treated patients with R5 HIV-1 infection. N Engl J Med. 2008 Oct 2;359(14):1429-41. doi: 10.1056/NEJMoa0803152. PMID 18832244
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001027&StudyName=Trial%20of%20Maraviroc%20%28UK-427%2C857%29%20in%20Combination%20with%20Optimized%20Background%20Therapy%20Versus%20Optimized%20Background%20Therapy%20Alone%20for%20the%20Tre

RESULTS

PARTICIPANT FLOW:
Groups:
- Maraviroc QD, Double Blind: Maraviroc 150 or 300 milligrams (mg) tablet orally once daily (QD) in the evening, dose adjusted according to the other prescribed drugs taken by participants as part of optimized background therapy (OBT) selected according to local standard of care (3 to 6 drugs based on resistance testing, treatment history and safety considerations). Placebo matched to maraviroc tablet orally in the morning.
- Maraviroc BID, Double Blind: Maraviroc 150 or 300 mg tablet orally twice daily (BID) in the morning and evening, dose adjusted according to the other prescribed drugs taken by participants as part of OBT selected according to local standard of care (3 to 6 drugs based on resistance testing, treatment history and safety considerations).
- Placebo, Double Blind: Placebo matched to maraviroc tablet orally BID in the morning and evening, in combination with OBT selected according to local standard of care (3 to 6 drugs based on resistance testing, treatment history and safety considerations).
- Maraviroc BID, Open Label: Participants from maraviroc QD, maraviroc BID and Placebo (double blind phase) who received maraviroc 150 or 300 mg BID in the morning and evening, dose adjusted according to the other prescribed drugs taken by participants as part of OBT selected according to local standard of care (3 to 6 drugs based on resistance testing, treatment history and safety considerations) during open label phase.
- In Study-off Drug (ISOD), Open Label: Participants from maraviroc QD, maraviroc BID and Placebo (double blind phase) who received no study treatment along with OBT selected according to local standard of care (3 to 6 drugs based on resistance testing, treatment history and safety considerations) in during open label phase.
- Maraviroc BID, Observation Phase: Participants continuing from open label phase, who received maraviroc 150 or 300 mg BID in the morning and evening, dose adjusted according to the other prescribed drugs taken by participants as part of OBT selected according to local standard of care (3 to 6 drugs based on resistance testing, treatment history and safety considerations) during observational phase.
- In Study-off Drug (ISOD), Observation Phase: Participants continuing from open label phase, who received no study treatment along with OBT selected according to local standard of care (3 to 6 drugs based on resistance testing, treatment history and safety considerations) during observational phase.
Period: Double Blind
Arm/Group | Maraviroc QD, Double Blind | Maraviroc BID, Double Blind | Placebo, Double Blind | Maraviroc BID, Open Label | In Study-off Drug (ISOD), Open Label | Maraviroc BID, Observation Phase | In Study-off Drug (ISOD), Observation Phase
Started | 241 | 240 | 120 | 0 | 0 | 0 | 0
Treated | 232 | 235 | 118 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 241 | 240 | 120 | 0 | 0 | 0 | 0
Not completed — Randomized, not treated | 9 | 5 | 2 | 0 | 0 | 0 | 0
Not completed — Ongoing at cut-off date | 151 | 166 | 72 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 11 | 10 | 6 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 43 | 34 | 17 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 4 | 1 | 0 | 0 | 0 | 0
Not completed — Participant defaulted | 19 | 18 | 11 | 0 | 0 | 0 | 0
Not completed — Un-specified | 7 | 3 | 11 | 0 | 0 | 0 | 0
Period: Open Label
Arm/Group | Maraviroc QD, Double Blind | Maraviroc BID, Double Blind | Placebo, Double Blind | Maraviroc BID, Open Label | In Study-off Drug (ISOD), Open Label | Maraviroc BID, Observation Phase | In Study-off Drug (ISOD), Observation Phase
Started | 0 | 0 | 0 | 327 | 62 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 327 | 62 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 13 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 4 | 0 | 0 | 0
Not completed — Participant defaulted | 0 | 0 | 0 | 24 | 0 | 0 | 0
Not completed — Un-specified | 0 | 0 | 0 | 15 | 0 | 0 | 0
Not completed — Ongoing at cut-off date | 0 | 0 | 0 | 269 | 62 | 0 | 0
Period: Observational Phase
Arm/Group | Maraviroc QD, Double Blind | Maraviroc BID, Double Blind | Placebo, Double Blind | Maraviroc BID, Open Label | In Study-off Drug (ISOD), Open Label | Maraviroc BID, Observation Phase | In Study-off Drug (ISOD), Observation Phase
Started | 0 | 0 | 0 | 0 | 0 | 250 | 81
Completed | 0 | 0 | 0 | 0 | 0 | 204 | 55
Not Completed | 0 | 0 | 0 | 0 | 0 | 46 | 26
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 5 | 4
Not completed — Participant defaulted | 0 | 0 | 0 | 0 | 0 | 34 | 18
Not completed — Un-specified | 0 | 0 | 0 | 0 | 0 | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Maraviroc QD: Maraviroc 150 or 300 milligrams (mg) tablet orally once daily (QD) in the evening, dose adjusted according to the other prescribed drugs taken by participants as part of optimized background therapy (OBT) selected according to local standard of care (3 to 6 drugs based on resistance testing, treatment history and safety considerations). Placebo matched to maraviroc tablet orally in the morning.
- Maraviroc BID: Maraviroc 150 or 300 mg tablet orally twice daily (BID) in the morning and evening, dose adjusted according to the other prescribed drugs taken by participants as part of OBT selected according to local standard of care (3 to 6 drugs based on resistance testing, treatment history and safety considerations).
- Placebo: Placebo matched to maraviroc tablet orally BID in the morning and evening, in combination with OBT (3 to 6 drugs based on resistance testing, treatment history and safety considerations).
- Total: Total of all reporting groups
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo | Total
Number analyzed (Participants) | 232 | 235 | 118 | 585
Age, Customized [Number; unit: participants] — Out of a total of 601 participants, data for baseline measure (age) was available for 585 participants who were treated.
  participants
    Less than 18 years | 0 | 0 | 0 | 0
    18 to 24 years | 1 | 0 | 0 | 1
    25 to 34 years | 10 | 7 | 5 | 22
    35 to 44 years | 97 | 108 | 48 | 253
    45 to 54 years | 93 | 90 | 45 | 228
    55 to 64 years | 26 | 28 | 19 | 73
    Greater than or equal to 65 years | 5 | 2 | 1 | 8
Sex: Female, Male [Count of Participants; unit: Participants] — Out of a total of 601 participants, data for baseline measure (gender) was available for 585 participants who were treated.
  Participants
    Female | 22 | 23 | 12 | 57
    Male | 210 | 212 | 106 | 528

OUTCOME MEASURES:

1. Primary Outcome: Log 10-transformed Human Immunodeficiency Virus Ribonucleic Acid (HIV-1 RNA) Levels at Baseline
Description: Baseline value calculated as average of pre-dose measurements collected at screening, randomization, and immediately pre-dose.
Time Frame: Baseline
Population: Full analysis set (FAS) included all the randomized participants who had taken at least one dose of the study medication.
Measure: Mean (Standard Deviation); unit: log10 copies/milliliter(log10 copies/mL)
Groups:
- Placebo: Placebo matched to maraviroc tablet orally BID in the morning and evening, in combination with OBT selected according to local standard of care (3 to 6 drugs based on resistance testing, treatment history and safety considerations).
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 232 | 235 | 118
log10 copies/milliliter(log10 copies/mL) | 4.854 (0.641) | 4.861 (0.614) | 4.840 (0.556)

2. Primary Outcome: Change From Baseline in Log 10-transformed HIV-1 RNA Levels at Week 24
Description: Change from baseline in log 10-transformed plasma viral load (HIV-1 RNA) levels (log10 copies/mL). Baseline value calculated as average of pre-dose measurements collected at screening, randomization, and immediately pre-dose.
Time Frame: Baseline and Week 24
Population: FAS included all the randomized participants who had taken at least one dose of the study medication. Missing values for viral load at week 24 have been imputed as baseline value for the participants who discontinued and as Last observation carried forward (LOCF) for participants who did not discontinue.
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 232 | 235 | 118
log10 copies/mL | -1.818 (0.0920) | -1.952 (0.0913) | -1.030 (0.1287)
Statistical Analysis 1: Comparison: Maraviroc QD vs Placebo; The difference between the treatment least square means (LS means) adjusted for the randomization strata was presented in addition to 2-sided 97.5% confidence interval (CI) as an adjustment for multiplicity using a Bonferroni correction. Negative value favors maraviroc over placebo; Test type: Superiority or Other; LS mean difference = -0.788, 97.5% CI 2-sided [-1.141 to -0.435], Standard Error of Mean 0.1571
Statistical Analysis 2: Comparison: Maraviroc BID vs Placebo; The difference between the treatment LS means adjusted for the randomization strata was presented in addition to 2-sided 97.5% CI as an adjustment for multiplicity using a Bonferroni correction. Negative value favors maraviroc over placebo; Test type: Superiority or Other; LS mean difference = -0.922, 97.5% CI 2-sided [-1.275 to -0.570], Standard Error of Mean 0.1568

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA Levels Less Than 400 Copies/mL
Time Frame: Week 24 and 48
Population: FAS included all the randomized participants who had taken at least one dose of the study medication. Missing data was imputed as "failure" which was defined as not meeting the criteria of less than 400 copies/mL of HIV-1 RNA levels.
Measure: Number; unit: percentage of participants
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 232 | 235 | 118
percentage of participants
  Week 24 | 54.7 | 60.4 | 31.4
  Week 48 | 50.9 | 57.5 | 22.0
Statistical Analysis 1: Comparison: Maraviroc QD vs Placebo; Week 24: Two-sided 95% CI was presented for the odds ratios between treatment groups with placebo as the comparator. CIs were calculated using the Wald-approximation. Logistic model with treatment, screening HIV concentrations (less than [<] 100,000 or greater than or equal to [>=] 100,000), enfuvirtide use (Yes or No) as covariates was used. Odds ratio greater than (>) 1 favors maraviroc; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.88, 95% CI 2-sided [1.78 to 4.67]
Statistical Analysis 2: Comparison: Maraviroc BID vs Placebo; Week 24: Two-sided 95% CI was presented for the odds ratios between treatment groups with placebo as the comparator. CIs were calculated using the Wald-approximation. Logistic model with treatment, screening HIV concentrations (<100,000 or >=100,000), enfuvirtide use (Yes or No) as covariates was used. Odds ratio >1 favors maraviroc; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.66, 95% CI 2-sided [2.26 to 5.95]
Statistical Analysis 3: Comparison: Maraviroc QD vs Placebo; Week 48: Two-sided 95% CI was presented for the odds ratios between treatment groups with placebo as the comparator. CIs were calculated using the Wald-approximation. Logistic model with treatment, screening HIV concentrations (<100,000 or >=100,000), enfuvirtide use (Yes or No) as covariates was used. Odds ratio >1 favors maraviroc; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.96, 95% CI 2-sided [2.36 to 6.64]
Statistical Analysis 4: Comparison: Maraviroc BID vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 5.11, 95% CI 2-sided [3.04 to 8.59]

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA Levels Less Than 400 Copies/mL or With at Least 0.5 log10 Decrease From Baseline
Time Frame: Week 24 and 48
Population: FAS included all the randomized participants who had taken at least one dose of the study medication. Missing data was imputed as "failure" which was defined as not meeting the criteria of less than 400 copies/mL or with at least 0.5 log10 decrease from baseline of HIV-1 RNA levels.
Measure: Number; unit: percentage of participants
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 232 | 235 | 118
percentage of participants
  Week 24 | 67.7 | 69.4 | 45.8
  Week 48 | 59.9 | 64.3 | 35.6
Statistical Analysis 1: Comparison: Maraviroc QD vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.60, 95% CI 2-sided [1.63 to 4.13]
Statistical Analysis 2: Comparison: Maraviroc BID vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.85, 95% CI 2-sided [1.79 to 4.54]
Statistical Analysis 3: Comparison: Maraviroc QD vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.93, 95% CI 2-sided [1.83 to 4.67]
Statistical Analysis 4: Comparison: Maraviroc BID vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.33, 95% CI 2-sided [2.08 to 5.32]

5. Secondary Outcome: Percentage of Participants With HIV-1 RNA Levels Less Than 400 Copies/mL or With at Least 1.0 log10 Decrease From Baseline
Time Frame: Week 24 and 48
Population: FAS included all the randomized participants who had taken at least one dose of the study medication. Missing data was imputed as "failure" which was defined as not meeting the criteria of less than 400 copies/mL or with at least 1.0 log10 decrease from baseline of HIV-1 RNA levels.
Measure: Number; unit: percentage of participants
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 232 | 235 | 118
percentage of participants
  Week 24 | 64.7 | 67.7 | 38.1
  Week 48 | 57.8 | 63.0 | 31.4
Statistical Analysis 1: Comparison: Maraviroc QD vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.06, 95% CI 2-sided [1.92 to 4.88]
Statistical Analysis 2: Comparison: Maraviroc BID vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.55, 95% CI 2-sided [2.22 to 5.68]
Statistical Analysis 3: Comparison: Maraviroc QD vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.30, 95% CI 2-sided [2.05 to 5.31]
Statistical Analysis 4: Comparison: Maraviroc BID vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.03, 95% CI 2-sided [2.50 to 6.51]

6. Secondary Outcome: Percentage of Participants With HIV-1 RNA Levels Less Than 50 Copies/mL
Time Frame: Week 24 and 48
Population: FAS included all the randomized participants who had taken at least one dose of the study medication. Missing data was imputed as "failure" which was defined as not meeting the criteria of less than 50 copies/mL of HIV-1 RNA levels.
Measure: Number; unit: percentage of participants
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 232 | 235 | 118
percentage of participants
  Week 24 | 42.2 | 48.5 | 24.6
  Week 48 | 41.8 | 46.8 | 16.1
Statistical Analysis 1: Comparison: Maraviroc QD vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 2.43, 95% CI 2-sided [1.46 to 4.04]
Statistical Analysis 2: Comparison: Maraviroc BID vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.15, 95% CI 2-sided [1.90 to 5.23]
Statistical Analysis 3: Comparison: Maraviroc QD vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.10, 95% CI 2-sided [2.32 to 7.25]
Statistical Analysis 4: Comparison: Maraviroc BID vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.97, 95% CI 2-sided [2.82 to 8.77]

7. Secondary Outcome: Cluster of Differentiation 4 (CD4) and Cluster of Differentiation 8 (CD8) Cell Count at Baseline
Description: Baseline value calculated as average of pre-dose measurements collected at screening and immediately pre-dose.
Time Frame: Baseline
Population: FAS included all the randomized participants who had taken at least one dose of the study medication. 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: cells per microliter (cells/µL)
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 231 | 235 | 118
cells per microliter (cells/µL)
  CD4 | 187.5 (149.88) | 176.5 (143.93) | 178.5 (127.09)
  CD8 | 941.1 (556.53) | 880.1 (547.19) | 880.4 (489.28)

8. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 24 and 48
Description: Change from baseline in CD4 cell count measured as cells/µL. Baseline value calculated as the average of pre-dose measurements collected at screening and immediately pre-dose.
Time Frame: Baseline, Week 24 and 48
Population: FAS included all the randomized participants who had taken at least one dose of the study medication. 'N' (number of participants analyzed) signifies participants evaluable for this measure. Missing values were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: cells/µL
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 227 | 233 | 116
cells/µL
  Week 24 | 106.63 (7.255) | 111.08 (7.148) | 52.14 (10.140)
  Week 48 | 112.53 (7.390) | 122.44 (7.284) | 53.97 (10.341)
Statistical Analysis 1: Comparison: Maraviroc QD vs Placebo; Week 24: The difference between the treatment LS means adjusted for the randomization strata was presented in addition to 2-sided 95% CI. Positive value favors maraviroc over placebo; Test type: Superiority or Other; LS mean difference = 54.49, 95% CI 2-sided [30.07 to 78.92], Standard Error of Mean 12.435
Statistical Analysis 2: Comparison: Maraviroc BID vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; LS mean difference = 58.94, 95% CI 2-sided [34.63 to 83.26], Standard Error of Mean 12.378
Statistical Analysis 3: Comparison: Maraviroc QD vs Placebo; Week 48: The difference between the treatment LS means adjusted for the randomization strata was presented in addition to 2-sided 95% CI. Positive value favors maraviroc over placebo; Test type: Superiority or Other; LS mean difference = 58.56, 95% CI 2-sided [33.66 to 83.46], Standard Error of Mean 12.677
Statistical Analysis 4: Comparison: Maraviroc BID vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority or Other; LS mean difference = 68.47, 95% CI 2-sided [43.69 to 93.25], Standard Error of Mean 12.617

9. Secondary Outcome: Change From Baseline in CD8 Cell Count at Week 24 and 48
Description: Change from baseline in CD8 cell count measured as cells/µL. Baseline value calculated as the average of pre-dose measurements collected at screening and immediately pre-dose.
Time Frame: Baseline, Week 24 and 48
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: cells/µL
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 227 | 233 | 116
cells/µL
  Week 24 | 283.48 (30.206) | 302.33 (29.745) | -0.74 (42.198)
  Week 48 | 198.00 (28.962) | 220.40 (28.532) | -15.34 (40.503)
Statistical Analysis 1: Comparison: Maraviroc QD vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; LS mean difference = 284.21, 95% CI 2-sided [182.51 to 385.92], Standard Error of Mean 51.779
Statistical Analysis 2: Comparison: Maraviroc BID vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; LS mean difference = 303.07, 95% CI 2-sided [201.90 to 404.23], Standard Error of Mean 51.507
Statistical Analysis 3: Comparison: Maraviroc QD vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority or Other; LS mean difference = 213.34, 95% CI 2-sided [115.77 to 310.92], Standard Error of Mean 49.679
Statistical Analysis 4: Comparison: Maraviroc BID vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority or Other; LS mean difference = 235.74, 95% CI 2-sided [138.68 to 332.80], Standard Error of Mean 49.416

10. Secondary Outcome: Time to Virological Failure
Description: Time to virologic failure based on observed HIV-1 RNA levels and failure events (death;permanent discontinuation of drug;lost to follow-up [LTFU];new anti-retroviral drug added [except background drug change to drug of same class];or on open label for early non-response or rebound). Failure:at Time 0 if level not <400 copies/mL(2 consecutive visits) before events or last available visit;at time of earliest event if level <400 copies/mL(2 consecutive visits);failure if level >=400 copies/mL(2 consecutive visits) or 1 visit >=400 copies/mL followed by permanent discontinuation of drug or LTFU.
Time Frame: Week 48
Population: FAS included all the randomized participants who had taken at least one dose of the study medication.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 232 | 235 | 118
days | 344.00 [195.00 to 372.00] | NA [NA to NA] — Data was not estimable because less than 50% of participants experienced virological failure. | 0.00 [NA to NA] — Data was not estimable because the empirical distribution of the data rendered the algorithmic formula non-calculable.
Statistical Analysis 1: Comparison: Maraviroc QD vs Placebo; P-value was calculated using Log rank test controlling for the effect of the randomization strata. Hazard ratio calculated by fitting a Cox proportional hazards model including treatment group and randomization strata. Hazard ratio <1 favors maraviroc; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.34 to 0.60]
Statistical Analysis 2: Comparison: Maraviroc BID vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.38, 95% CI 2-sided [0.28 to 0.50]

11. Secondary Outcome: Time-Averaged Difference (TAD) From Baseline in log10 Transformed HIV-1 RNA Levels
Description: TAD from baseline was calculated as area under the curve of HIV-1 RNA load (log10 copies/mL) divided by time period minus baseline HIV-1 RNA load (log10 copies/mL). Baseline value calculated as the average of pre-dose measurements collected at screening, randomization, and immediately pre-dose.
Time Frame: Baseline to Week 24 and Week 48
Population: FAS included all the randomized participants who had taken at least one dose of the study medication. Missing data imputed as 0 for participants who discontinued and through last available observation for participants who did not discontinue.
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 232 | 235 | 118
log10 copies/mL
  Week 24 | -1.636 (0.0789) | -1.741 (0.0783) | -0.939 (0.1103)
  Week 48 | -1.556 (0.0876) | -1.720 (0.0870) | -0.788 (0.1227)
Statistical Analysis 1: Comparison: Maraviroc QD vs Placebo; Week 24: The difference between the treatment LS means adjusted for the randomization strata was presented in addition to 2-sided 95% CI. Negative value favors maraviroc over placebo; Test type: Superiority or Other; LS mean difference = -0.697, 95% CI 2-sided [-0.961 to -0.432], Standard Error of Mean 0.1347
Statistical Analysis 2: Comparison: Maraviroc BID vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; LS mean difference = -0.802, 95% CI 2-sided [-1.065 to -0.538], Standard Error of Mean 0.1344
Statistical Analysis 3: Comparison: Maraviroc QD vs Placebo; Week 48: The difference between the treatment LS means adjusted for the randomization strata was presented in addition to 2-sided 95% CI. Negative value favors maraviroc over placebo; Test type: Superiority or Other; LS mean difference = -0.767, 95% CI 2-sided [-1.061 to -0.474], Standard Error of Mean 0.1497
Statistical Analysis 4: Comparison: Maraviroc BID vs Placebo; [analysis description as in outcome 11, analysis 3]; Test type: Superiority or Other; LS mean difference = -0.931, 95% CI 2-sided [-1.225 to -0.638], Standard Error of Mean 0.1494

12. Primary Outcome: Change From Baseline in Log 10-transformed HIV-1 RNA Levels at Week 48
Description: Change from baseline in log 10-transformed plasma viral load (HIV-1 RNA) levels (log10 copies/mL). Baseline value calculated as average of pre-dose measurements collected at screening, randomization and immediately pre-dose.
Time Frame: Baseline and Week 48
Population: FAS included all the randomized participants who had taken at least one dose of the study medication. Missing values for viral load at week 48 have been imputed as the baseline value for participants who discontinued and as LOCF for participants who did not discontinue.
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 232 | 235 | 118
log10 copies/mL | -1.656 (0.0949) | -1.824 (0.0942) | -0.803 (0.1329)
Statistical Analysis 1: Comparison: Maraviroc QD vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -0.853, 97.5% CI 2-sided [-1.217 to -0.489], Standard Error of Mean 0.1621
Statistical Analysis 2: Comparison: Maraviroc BID vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -1.021, 97.5% CI 2-sided [-1.385 to -0.658], Standard Error of Mean 0.1618

13. Secondary Outcome: Number of Participants With Genotypic Susceptibility Scores (GSS) and Phenotypic Susceptibility Score (PSS) at Screening
Description: Number of participants with GSS and PSS were used as surrogates for assessing genotype and phenotype. Genotypic and phenotypic resistance to protease inhibitors(PIs), nucleoside reverse transcriptase inhibitors(NRTIs), non-nucleoside reverse transcriptase inhibitors(NNRTIs) were evaluated at screening (not at baseline), by Monogram Biosciences PhenoSense genotyping (GT) assay. Score was determined for each drug in OBT, giving 1:drug 'sensitive'/'susceptible' and 0:'resistant'. GSS and PSS score range:0 to >3. Genotypic enfuvirtide value was used for PSS, no phenotypic enfuvirtide was recorded.
Time Frame: Screening
Population: FAS included all the randomized participants who had taken at least one dose of the study medication.
Measure: Number; unit: participants
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 232 | 235 | 118
participants
  GSS: 0 | 52 | 59 | 31
  GSS: 1 | 82 | 80 | 29
  GSS: 2 | 38 | 48 | 21
  GSS: greater than or equal to 3 | 57 | 47 | 34
  GSS: missing | 3 | 1 | 3
  PSS: 0 | 25 | 24 | 17
  PSS: 1 | 70 | 73 | 18
  PSS: 2 | 51 | 69 | 35
  PSS: greater than or equal to 3 | 83 | 66 | 45
  PSS: missing | 3 | 3 | 3

14. Secondary Outcome: Number of Participants With Change in GSS and PSS From Screening at the Time of Treatment Failure Through Week 24
Description: Number of participants with GSS and PSS were used as surrogates for assessing genotype and phenotype. Genotypic and phenotypic resistance to PIs, NRTIs and NNRTIs were evaluated at screening and time of treatment failure analyzed through week 24 visit, by Monogram Biosciences PhenoSense GT assay. Score was determined for each drug in OBT, giving 1: drug 'sensitive'/'susceptible' and 0: 'resistant'. GSS and PSS score range:0 to >3. Genotypic enfuvirtide value was used for PSS, no phenotypic enfuvirtide was recorded.
Time Frame: Screening and time of failure through week 24
Population: FAS; 'N' (number of participants analyzed) is signifying those participants who experienced treatment failure defined as discontinuation due to insufficient response. 'n' is number of participants who were evaluable for the given change in GSS and PSS score for each arm group respectively.
Measure: Number; unit: participants
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 42 | 46 | 53
participants
  Change in GSS by less than -3 (n= 35 ,40, 47) | 0 | 0 | 1
  Change in GSS by -3 (n= 35 ,40, 47) | 0 | 0 | 0
  Change in GSS by -2 (n= 35 ,40, 47) | 3 | 0 | 1
  Change in GSS by -1 (n= 35 ,40, 47) | 9 | 13 | 11
  Change in GSS by 0 (n= 35 ,40, 47) | 23 | 26 | 32
  Change in GSS by 1 (n= 35 ,40, 47) | 0 | 1 | 1
  Change in GSS by 2 (n= 35 ,40, 47) | 0 | 0 | 0
  Change in GSS by 3 (n= 35 ,40, 47) | 0 | 0 | 1
  Change in GSS by greater than 3 (n= 35 ,40, 47) | 0 | 0 | 0
  Change in PSS by less than -3 (n= 35 ,40, 45) | 0 | 0 | 1
  Change in PSS by -3 (n= 35 ,40, 45) | 4 | 1 | 1
  Change in PSS by -2 (n= 35 ,40, 45) | 4 | 1 | 4
  Change in PSS by -1 (n= 35 ,40, 45) | 10 | 18 | 12
  Change in PSS by 0 (n= 35 ,40, 45) | 15 | 17 | 25
  Change in PSS by 1 (n= 35 ,40, 45) | 2 | 3 | 2
  Change in PSS by 2 (n= 35 ,40, 45) | 0 | 0 | 0
  Change in PSS by 3 (n= 35 ,40, 45) | 0 | 0 | 0
  Change in PSS by greater than 3 (n= 35 ,40, 45) | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Change in GSS and PSS From Screening at the Time of Treatment Failure at Week 48
Description: Number of participants with GSS and PSS were used as surrogates for assessing genotype and phenotype. Genotypic and phenotypic resistance to PIs, NRTIs and NNRTIs were evaluated at screening and time of treatment failure analyzed through week 48 visit, by Monogram Biosciences PhenoSense GT assay. Score was determined for each drug in OBT, giving 1: drug 'sensitive'/'susceptible' and 0: 'resistant'. GSS and PSS score range:0 to >3. Genotypic enfuvirtide value was used for PSS, no phenotypic enfuvirtide was recorded.
Time Frame: Screening and time of failure through week 48
Population: FAS; 'N' (number of participants analyzed) is signifying those participants who experienced treatment failure defined as discontinuation due to discontinuation due to insufficient response. 'n' is number of participants who were evaluable for the given change in GSS and PSS score for each arm group respectively.
Measure: Number; unit: participants
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 51 | 58 | 62
participants
  Change in GSS by less than -3 (n= 44 ,52, 55) | 0 | 0 | 1
  Change in GSS by -3 (n= 44 ,52, 55) | 0 | 0 | 1
  Change in GSS by -2 (n= 44 ,52, 55) | 5 | 1 | 2
  Change in GSS by -1 (n= 44 ,52, 55) | 12 | 17 | 15
  Change in GSS by 0 (n= 44 ,52, 55) | 26 | 31 | 33
  Change in GSS by 1 (n= 44 ,52, 55) | 1 | 2 | 1
  Change in GSS by 2 (n= 44 ,52, 55) | 0 | 1 | 1
  Change in GSS by 3 (n= 44 ,52, 55) | 0 | 0 | 1
  Change in GSS by greater than 3 (n= 44 ,52, 55) | 0 | 0 | 0
  Change in PSS by less than -3 (n= 44 , 52, 53) | 0 | 1 | 1
  Change in PSS by -3 (n= 44 , 52, 53) | 4 | 1 | 3
  Change in PSS by -2 (n= 44 , 52, 53) | 6 | 3 | 6
  Change in PSS by -1 (n= 44 , 52, 53) | 13 | 21 | 12
  Change in PSS by 0 (n= 44 , 52, 53) | 17 | 23 | 26
  Change in PSS by 1 (n= 44 , 52, 53) | 3 | 3 | 4
  Change in PSS by 2 (n= 44 , 52, 53) | 0 | 0 | 1
  Change in PSS by 3 (n= 44 , 52, 53) | 1 | 0 | 0
  Change in PSS by greater than 3 (n= 44 , 52, 53) | 0 | 0 | 0

16. Secondary Outcome: Number of Participants Per Tropism Status at Baseline and at the Time of Treatment Failure Through Week 24
Description: Number of participants per tropism status (C-X-C chemokine receptor 5 {CCR5} [R5], C-X-C chemokine receptor type 4 {CXCR4} [X4], Dual/mixed [DM], or Non-reportable/Non-phenotypable [NR/NP]) at baseline and time of treatment failure analyzed through week 24 visit. Treatment failure defined as discontinuation due to insufficient clinical response. HIV-1 RNA viral load <500 copies/mL categorized as below lower limit of quantification (BLQ). The assessment for time of treatment failure was defined as the last on treatment assessment.
Time Frame: Baseline and time of failure through week 24
Population: FAS; 'N' (number of participants analyzed) is signifying those participants who experienced treatment failure, defined as discontinuation due to insufficient response and had tropism assessment at baseline.
Measure: Number; unit: participants
Groups:
- Maraviroc QD: Description Maraviroc 150 or 300 milligrams (mg) tablet orally once daily (QD) in the evening, dose adjusted according to the other prescribed drugs taken by participants as part of optimized background therapy (OBT) selected according to local standard of care (3 to 6 drugs based on resistance testing, treatment history and safety considerations). Placebo matched to maraviroc tablet orally in the morning.
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 42 | 46 | 53
participants
  Baseline: R5; Treatment failure: R5 | 10 | 10 | 44
  Baseline: R5; Treatment failure: X4 | 6 | 5 | 0
  Baseline: R5; Treatment failure: DM | 18 | 19 | 1
  Baseline: R5; Treatment failure: NR/NP | 1 | 3 | 3
  Baseline: DM; Treatment failure: R5 | 0 | 0 | 1
  Baseline: DM; Treatment failure: X4 | 1 | 4 | 1
  Baseline: DM; Treatment failure: DM | 3 | 4 | 1
  Baseline: DM; Treatment failure: NR/NP | 1 | 1 | 0

17. Secondary Outcome: Number of Participants Per Tropism Status at Baseline and at the Time of Treatment Failure Through Week 48
Description: Number of participants per tropism status (R5, X4, DM, or NR/NP) at baseline and time of treatment failure analyzed through week 48 visit. Treatment failure defined as insufficient clinical response. HIV-1 RNA viral load <500 copies/mL categorized as BLQ. The assessment for time of treatment failure was defined as the last on treatment assessment.
Time Frame: Baseline and time of failure through week 48
Population: as for outcome 16
Measure: Number; unit: participants
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 51 | 58 | 62
participants
  Baseline: R5, Treatment failure: R5 | 16 | 15 | 49
  Baseline: R5, Treatment failure: X4 | 6 | 7 | 0
  Baseline: R5, Treatment failure: DM | 19 | 22 | 3
  Baseline: R5, Treatment failure: NR/NP | 1 | 3 | 3
  Baseline: DM, Treatment failure: R5 | 0 | 0 | 2
  Baseline: DM, Treatment failure: X4 | 2 | 4 | 1
  Baseline: DM, Treatment failure: DM | 4 | 5 | 1
  Baseline: DM, Treatment failure: NR/NP | 2 | 1 | 0

18. Secondary Outcome: Change From Baseline in Viral Load at Week 24 and Week 48 by Overall Susceptibility Score (OSS) at Screening
Description: Association between baseline resistance and virological response was assessed as change in viral load by OSS at screening. OSS categorized as 0, 1, 2, >3 (maximum value of 6) and calculated as the sum of the net assessment of in-vitro phenotypic and genotypic susceptibility using a binary scoring system (0= resistant, 1= sensitive or susceptible) for each antiretroviral agent in OBT. Higher scores indicate greater susceptibility. Baseline value is the average of the values from screening, randomization and immediately pre-dose.
Time Frame: Baseline, Week 24 and Week 48
Population: FAS; 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure. 'n' is number of participants with given OSS score at screening for each treatment arm at particular time-point. LOCF was used to impute missing values.
Measure: Mean (Standard Deviation); unit: log10copies/mL
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 228 | 234 | 116
log10copies/mL
  Week 24; Screening OSS 0 (n= 29, 27, 19) | -0.945 (0.905) | -1.524 (1.331) | -0.083 (0.472)
  Week 24; Screening OSS 1 (n= 76, 86, 21) | -1.911 (1.229) | -1.895 (1.395) | -0.350 (0.784)
  Week 24; Screening OSS 2 (n= 51, 65, 38) | -2.093 (1.3402) | -2.220 (1.0900) | -1.251 (1.0800)
  Week 24; Screening OSS >=3 (n= 68, 53, 35) | -2.536 (1.1599) | -2.672 (1.1836) | -2.471 (0.9200)
  Week 24; Screening OSS= Missing (n= 4, 3, 3) | -2.070 (1.3832) | -3.075 (0.5705) | -0.530 (0.1726)
  Week 48; Screening OSS 0 (n= 29, 27, 19) | -0.876 (0.8448) | -1.419 (1.3042) | -0.088 (0.4541)
  Week 48; Screening OSS 1 (n= 77, 86, 20) | -1.843 (1.2452) | -1.868 (1.4078) | -0.262 (0.7048)
  Week 48; Screening OSS 2 (n= 51, 64, 38) | -2.146 (1.4208) | -2.182 (1.1096) | -1.147 (0.9681)
  Week 48; Screening OSS >=3 (n= 67, 54, 36) | -2.427 (1.3136) | -2.634 (1.1628) | -2.205 (1.0870)
  Week 48; Screening OSS= Missing (n= 4, 3, 3) | -2.106 (1.4461) | -2.698 (1.2056) | -0.370 (0.1471)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Maraviroc QD, Double Blind | Maraviroc BID, Double Blind | Placebo, Double Blind | Maraviroc BID, Open Label | In Study-off Drug (ISOD), Open Label | Maraviroc BID, Observation Phase | In Study-off Drug (ISOD), Observation Phase
Serious Adverse Events (participants affected / at risk) | 42/232 | 53/235 | 20/118 | 33/327 | 0/62 | 0/250 | 0/81
Other Adverse Events (participants affected / at risk) | 170/232 | 192/235 | 89/118 | 19/327 | 0/62 | 0/250 | 0/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Maraviroc QD, Double Blind (N=232) | Maraviroc BID, Double Blind (N=235) | Placebo, Double Blind (N=118) | Maraviroc BID, Open Label (N=327) | In Study-off Drug (ISOD), Open Label (N=62) | Maraviroc BID, Observation Phase (N=250) | In Study-off Drug (ISOD), Observation Phase (N=81)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blindness unilateral (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 2 | 2 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 3 | 0 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 3 | 1 | 2 | 2 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 5 | 1 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Antiphospholipid syndrome (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthritis gonococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cavernous sinus thrombosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
HIV wasting syndrome (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infective myositis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0/0 | 0
Pneumonia (Infections and infestations) | 7 | 2 | 4 | 1 | 0 | 0 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Urethral abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
HIV infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mycobacterium avium complex infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nuclear magnetic resonance imaging brain (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint warmth (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 2 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1 | 2 | 0 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Sweat gland tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumocephalus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hip surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Plasmapheresis (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stent placement (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Toe operation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infarction (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc QD, Double Blind (N=232) | Maraviroc BID, Double Blind (N=235) | Placebo, Double Blind (N=118) | Maraviroc BID, Open Label (N=327) | In Study-off Drug (ISOD), Open Label (N=62) | Maraviroc BID, Observation Phase (N=250) | In Study-off Drug (ISOD), Observation Phase (N=81)
Abdominal distension (Gastrointestinal disorders) | 13 | 9 | 4 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 12 | 13 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 12 | 16 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 58 | 53 | 30 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 45 | 48 | 23 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 20 | 15 | 12 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 36 | 46 | 22 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 20 | 24 | 14 | 0 | 0 | 0 | 0
Malaise (General disorders) | 3 | 1 | 6 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 13 | 9 | 3 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 19 | 32 | 13 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 20 | 20 | 9 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 5 | 12 | 3 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 14 | 19 | 9 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 15 | 24 | 5 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 36 | 35 | 10 | 19 | 0 | 0 | 0
Weight decreased (Investigations) | 14 | 8 | 2 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 19 | 17 | 4 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 20 | 3 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 20 | 8 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 | 6 | 5 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 11 | 5 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 27 | 25 | 9 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 34 | 35 | 19 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 12 | 9 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 15 | 14 | 4 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 22 | 25 | 7 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 31 | 37 | 8 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 15 | 4 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 16 | 4 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 12 | 2 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 10 | 16 | 3 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 19 | 24 | 6 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 6 | 12 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.